CLINICAL TRIAL: NCT03141853
Title: Equine-assisted Therapy for Adults and Older Adults With Arthritis: A Randomized Controlled Trial
Brief Title: Horses and Education as Arthritis Therapy
Acronym: HEAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri, Kansas City (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16-276
Record Dates: First submitted 2017-03-20; First posted 2017-05-05 (Actual); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Arthritis
Keywords: Randomized Controlled Trial; Intervention Study
MeSH Terms: conditions — Arthritis | interventions — Equine-Assisted Therapy

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial. One group will receive equine-assisted therapy and the second group will receive arthritis exercise education
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants, care provider, and outcomes assessor will be masked as to which is the intervention and which is the control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Equine-assisted Therapy Group (Experimental): This group will interact and ride horses for 1 hour each week for 6 weeks. Horses will remain at a walk and an standard Therapeutic Riding curriculum will be used including safety, mounting, riding, tasks while riding, dismount, bonding with the horse.
  Interventions: Other: Equine-assisted Therapy
- Arthritis Exercise Education Group (Placebo Comparator): This group will receive exercise education that targets arthritis symptoms for 1 hour each week for 6 weeks. This will be based on the exercise education from the Arthritis foundation How-to Exercise With Arthritis. (n.d.).
  Interventions: Other: Arthritis Exercise Education

INTERVENTIONS:
Other: Equine-assisted Therapy — Participants will groom and ride horses. Horses will be kept at a walk with tasks such as serpentine, circles, and zig zags to complete. Stretching, and tasks like throwing a ball into a net from horseback will be completed
  Other Names: Hippotherapy; Therapeutic Horseback Riding
  Arms: Equine-assisted Therapy Group
Other: Arthritis Exercise Education — Standard of Care from the Arthritis Foundation - How-to Exercise With Arthritis. (n.d.). Retrieved April 18, 2016, from http://www.arthritis.org/living-with-arthritis/exercise/how-to). This intervention will consist of 6 -1 hour education sessions once a week on exercise to improve symptoms of arthritis
  Arms: Arthritis Exercise Education Group

SUMMARY:
A study will be conducted to assess if adults and older adults with arthritis who ride horses are able to move better, have less pain, enjoy nature more and have a better quality of life then people who go to class to learn about exercise. This is needed because adults with arthritis experience joint pain, stiffness, damage to their cartilage, and decreased range of motion in their hips, knees, shoulders, and back. This study will measure effects on patient's joints, pain, quality of life, muscle and cartilage before and after either arthritis exercise education or horse riding. Horses have unique movements that target joints without weight bearing and possibly show improvements without joint damage.

Twenty two subjects will be assigned to either the equine-assisted therapy (EAT) group or a group receiving exercise education for 1 hour each week for 6 weeks. Outcomes of pain, joint mobility and quality of life are measured at 0, 3 and 6 weeks. Enjoyment will be determined by a survey. Safety procedures include helmets, side walking attendants for balance, and controlled by a certified riding instructor at a certified riding center. Data will be gathered and reviewed, to assess the effects of EAT on arthritis.

DETAILED DESCRIPTION:
The purpose of the proposed research is to assess the feasibility, acceptability and effects of equine-assisted therapy on adults and older adults with arthritis. Equine-assisted therapy (EAT) is defined as any intervention using the unique qualities of horses to improve social, gross motor, and self-help skills.(Ratliffe & Sanekane, 2009) Although equine therapy has been used as a medical intervention since the second century (Ratliffe & Sanekane, 2009), no research has been conducted using equine-assisted therapy to improve arthritis.

In the United States arthritis accounts for $128 billion in lost income and medical costs (Centers for Disease Control and Prevention (CDC), 2013) Incidence of arthritis is increasing due to obesity and an aging population.(Bijlsma, Berenbaum, & Lafeber, 2011) Adults aged 40 to 65 and older than 65 with arthritis experience joint pain, stiffness, damage to cartilage, and decreased range of motion particularly in hips, knees, shoulders, and back (Barten et al., 2015; George et al., 2015; Karjalainen et al., 2001). Practice recommendations of non-pharmacological management of arthritis include using a biopsychosocial approach, an individualized exercise regime, strengthening leg and hip muscles, and improving the range of motion for muscle and joint health (Fernandes et al., 2013). Healthy People 2020 reports that arthritis has a major effect on a person's quality of life, ability to work and activities of daily life with the objectives of decreasing joint pain, decrease limitations, and decreasing psychological stress. Improving arthritis includes decreasing pain and improving the arthritic impact on the individual's quality of life.(Buchbinder, Bombardier, Yeung, & Tugwell, 1995) To improve musculoskeletal and functional health, the (World Health Organization, 2010) recommends physical activity including aerobic physical activity, strength, flexibility and balance. Current treatments include the use of physical conditioning (Schaafsma et al., 2013), opioids (Chaparro et al., 2013), and injections of anti-inflammatory medications, morphine, anesthetics or steroids(Staal, de Bie, De Vet, Hildebrandt, & Nelemans, 2008). The side effects from these medications can be bothersome, thus non-pharmacologic interventions must be further explored to improve adults and older adults with arthritis. Equine assisted therapy is a promising option since unique movements of the horse translate tri-rotational movements from the horse to the human (Selby & Smith-Osborne, 2013). This targets the spine and hip joints by non-weight bearing movement and has the potential to improve outcomes without joint damage.

There are both physical and psychosocial medical uses for equine assisted therapy. Previous meta-analyses of horses used to improve cerebral palsy in children, provide evidence to support the physical-neuromuscular connection and improvements in outcomes (Nimer & Lundahl, 2007; Pretty et al., 2007; Tseng, Chen, & Tam, 2013) reported significant improvement in total mood when riding horses. Anticipated implications for this research include improved range of motion, decreased pain, improved quality of life and enjoyment of nature. The bio-markers will assess the implications on cartilage and muscle to monitor improvement, destruction, or maintenance of both during equine-assisted therapy. If quality of life, enjoyment of nature and range of motion increase without muscle or cartilage destruction, then this would present evidence that EAT is a viable and desirable intervention and this will lead to further research for arthritis interventions including equines.

ELIGIBILITY:
Inclusion Criteria:

- Ages 45 and older

Joint pain inclusion will be considered with a mild [Mild pain (0-44)] to moderate pain level [Moderate pain (45-74 mm)] (Hawker, Mian, Kendzerska, & French, 2011) not completely relieved by medications.

Measured decreased range of motion by 20% (back, shoulder, knee and hip) and hip abduction wide enough to straddle a horse without discomfort.

Written physician's or advanced practice registered nurse's (APRN) clearance to ride a horse.

Ability to read and understand English as evidenced by the capacity to follow verbal and written directions at the screening interview.

Exclusion Criteria:

Self-reported: fear of horses.

Self reported allergies to horses.

Self reported osteoporosis.

Inability to abduct hips wide enough to straddle a horse comfortably.

Lack of transportation to the Therapeutic Riding Center.

Horse riding for the previous six months.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-05-20 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Attendance - Measured by number of participants attending each arm of the study | 0, 1, 2, 3, 4, 5, and week 6
  Data on attendance will be collected at 0 (screening), 1, 2, 3, 4, 5, and week 6. Tracking of de-identified will be measured. Data will be aggregated according to intervention vs. control group.
Recruitment - Data will be measured according to number of participants. | Prior to and including Week 1 of the study
  Participant data will include: : Identified, Approached, Screened, Consented, and attending week 1 of either intervention
Implementation - This will be measured by completed Protocol Impediment Form | Measured after week 6
  Each time a roadblock or difficulty in implementation occurs a Protocol Impediment Form will be completed. Data from these forms will be aggregated for reporting of findings from the study
Fidelity to the Protocol - This is measured by a researcher or research assistant observing with a protocol checklist. | 0, 1, 2, 3, 4, 5, and week 6
  Each time there is a Protocol Violation the researcher or Research Assistant will correct the violation and mark that is was corrected. Data will be aggregated and reported for protocol violations in each arm
Recruitment Procedure Sequence - This will be measured by number of participants | Week 0, 1
  Number of participants approached will be compared to number of participants who meet inclusion criteria and then start week 1.
Exclusion of Participants - This is measured by number of participants that meet exclusion criteria | Week 0
  Reasons for exclusion will be aggregated and reported
Attrition - This is measured by the number of participants enrolled vs. completion of the study | 0, 6 weeks
  Attrition rate will be calculated and reported
Completeness - This will be measured by number of Protocol Impediment incidences, Protocol violations noted on the Protocol checklists. | 0, 1, 2, 3, 4, 5, and week 6
  Incidents of incomplete protocol will be measured, calculated and aggregated by Protocol step
Timing - measured by minutes for each major protocol step | 0, 1, 2, 3, 4, 5, and 6 Weeks
  Planned time vs. actual time for protocol steps will be collected and aggregated.
Compliance - This will be measured by number of Protocol Violations due to refusal or inability to comply with the protocol | 0, 1, 2, 3, 4, 5, and 6 Weeks
  Protocol Violations will be categorized into researcher violations, participant violations, therapeutic riding instructor violations.
Missing Data - Missing data will be counted | 8 Weeks
  Missing data will be identified and counted.
Acceptability of the protocol - measured by Exit Survey Questionaire | 6 Weeks
  Open ended question will be administered upon exit of the study asking about acceptability of the study protocol for each arm
Continuing the intervention - Measured by self reported affirmative responses | 8 Weeks
  Do the study participants intend to continue the intervention after the end of the study? This will be asked at the end of the study and a follow-up phone call to assess if they continued will be made at 8 weeks. Data will be aggregated and reported.
Migration - Measured by number of requests to move from assigned groups | 0, 1, 2, 3, 4, 5, and 6 Weeks
  Do the participants stay in the assigned groups, e.g. not wanting to move from control group to treatment group? Note of any desire to change groups will be documented and counted. Data will be aggregated and reported.
Blinding - Measured by number of responses of participants checking if they were in the intervention or control group | 6 Weeks
  Do participants know that they are in the treatment group or control group at the end of the study? At the conclusion of the study this will be asked. Data will be aggregated and reported.
Length of Study Visits - Measured by number of responses on a Likert scale on Exit survey | 6 Weeks
  Do the participants feel the time spent per session is too long, too short, or just right? This will be asked at the conclusion of the study. Data will be aggregated and reported.
Length of Overall Study - Measured by number of responses on Exit survey Likert scale | 6 Weeks
  Do the participants feel the time spent in the study (6 weeks) was too long, too short or just right? This will be asked at the conclusion of the study. Data will be aggregated and reported.
Measurement - Measured by number of responses on Exit Survey - Yes/No | 6 Weeks
  Do the participants feel the measures were too extensive. This will be asked and measured at the conclusion of the study. Data will be aggregated and reported.
Study Improvement - Measured by comments for improvement | 6 Weeks
  Any other suggestions for improving the study. Responses for improvement will be asked, documented and collated for themes.

SECONDARY OUTCOMES:
Pain | 0, 3, and 6 Weeks
  What is the effect of an equine-assisted therapy intervention compared to an exercise attention-control intervention on pain in adults and older adults with arthritis? Visual Analog Pain Scale will be used to measure
Range of Motion | 0, 3, and 6 Weeks
  What is the effect of an equine-assisted therapy intervention compared to an exercise attention-control intervention on range of motion in adults and older adults with arthritis? Goniometer will measure joint range of motion
Serum Troponin | 0 and 6 Weeks
  What is the effect of an equine-assisted therapy intervention compared to an exercise attention-control intervention on serum troponin for muscle in adults and older adults with arthritis? Serum Troponin will be used to measure this.
Cartilage Oligomeric Matrix Protein (COMP) Biomarker | 0 and 6 Weeks
  What is the effect of an equine-assisted therapy intervention compared to an exercise attention-control intervention on Cartilage Oligomeric Matrix Protein biomarker for cartilage in adults and older adults with arthritis? Serum COMP will be measured
Quality of Life | 0, 3, and 6 Weeks
  What is the effect of an equine-assisted therapy intervention compared to an exercise attention-control intervention on quality of life in adults and older adults with arthritis? Arthritis Impact Measurement Scale 2 (AIMS 2) short-form will be used to measure this.
Enjoyment of Nature | 0, 3, and 6 Weeks
  What is the effect of an equine-assisted therapy intervention compared to an exercise attention-control intervention on enjoyment of nature in adults and older adults with arthritis? Environmental Attitudes Inventory Scale Sub-scale #1 will measure this.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia L Russell, PhD, Study Chair — University of Missouri, Kansas City
Locations (3):
- United States (3):
  - Due West Therapeutic Riding Center, Kansas City, Kansas
  - Kansas City Physician's Partners, Kansas City, Missouri
  - Saint Luke's College of Health Sciences, Kansas City, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aranda-Garcia S, Iricibar A, Planas A, Prat-Subiran JA, Angulo-Barroso RM. Comparative effects of horse exercise versus traditional exercise programs on gait, muscle strength, and body balance in healthy older adults. J Aging Phys Act. 2015 Jan;23(1):78-89. doi: 10.1123/japa.2012-0326. Epub 2014 Jan 14. PMID 24425454
- [Background] Araujo TB, Silva NA, Costa JN, Pereira MM, Safons MP. Effect of equine-assisted therapy on the postural balance of the elderly. Rev Bras Fisioter. 2011 Sep-Oct;15(5):414-9. doi: 10.1590/s1413-35552011005000027. Epub 2011 Oct 14. English, Portuguese. PMID 22002189
- [Background] Barten DJ, Swinkels LC, Dorsman SA, Dekker J, Veenhof C, de Bakker DH. Treatment of hip/knee osteoarthritis in Dutch general practice and physical therapy practice: an observational study. BMC Fam Pract. 2015 Jun 27;16:75. doi: 10.1186/s12875-015-0295-9. PMID 26116374
- [Background] Beil K, Hanes D. The influence of urban natural and built environments on physiological and psychological measures of stress--a pilot study. Int J Environ Res Public Health. 2013 Mar 26;10(4):1250-67. doi: 10.3390/ijerph10041250. PMID 23531491
- [Background] Beinotti F, Christofoletti G, Correia N, Borges G. Effects of horseback riding therapy on quality of life in patients post stroke. Top Stroke Rehabil. 2013 May-Jun;20(3):226-32. doi: 10.1310/tsr2003-226. PMID 23841970
- [Background] Beinotti F, Correia N, Christofoletti G, Borges G. Use of hippotherapy in gait training for hemiparetic post-stroke. Arq Neuropsiquiatr. 2010 Dec;68(6):908-13. doi: 10.1590/s0004-282x2010000600015. PMID 21243251
- [Background] Bijlsma JW, Berenbaum F, Lafeber FP. Osteoarthritis: an update with relevance for clinical practice. Lancet. 2011 Jun 18;377(9783):2115-26. doi: 10.1016/S0140-6736(11)60243-2. PMID 21684382
- [Background] Bizub AL, Joy A, Davidson L. "It's like being in another world": demonstrating the benefits of therapeutic horseback riding for individuals with psychiatric disability. Psychiatr Rehabil J. 2003 Spring;26(4):377-84. doi: 10.2975/26.2003.377.384. PMID 12739908
- [Background] Boonstra AM, Schiphorst Preuper HR, Reneman MF, Posthumus JB, Stewart RE. Reliability and validity of the visual analogue scale for disability in patients with chronic musculoskeletal pain. Int J Rehabil Res. 2008 Jun;31(2):165-9. doi: 10.1097/MRR.0b013e3282fc0f93. PMID 18467932
- [Background] Borioni N, Marinaro P, Celestini S, Del Sole F, Magro R, Zoppi D, Mattei F, Dall' Armi V, Mazzarella F, Cesario A, Bonassi S. Effect of equestrian therapy and onotherapy in physical and psycho-social performances of adults with intellectual disability: a preliminary study of evaluation tools based on the ICF classification. Disabil Rehabil. 2012;34(4):279-87. doi: 10.3109/09638288.2011.605919. Epub 2011 Oct 12. PMID 21988646
- [Background] Boswell, S., Gusowski, K., Kaiser, A., & Flachenecker, P. (2009). Hippotherapy in multiple sclerosis - results of a prospective, controlled, randomised and single-blind trial. Poster presentation.
- [Background] Brock, B.J, (1988). Effect of therapeutic horseback riding on physically disabled adults
- [Background] Buchbinder R, Bombardier C, Yeung M, Tugwell P. Which outcome measures should be used in rheumatoid arthritis clinical trials? Clinical and quality-of-life measures' responsiveness to treatment in a randomized controlled trial. Arthritis Rheum. 1995 Nov;38(11):1568-80. doi: 10.1002/art.1780381108. PMID 7488277
- [Background] Burch PM, Pogoryelova O, Goldstein R, Bennett D, Guglieri M, Straub V, Bushby K, Lochmuller H, Morris C. Muscle-Derived Proteins as Serum Biomarkers for Monitoring Disease Progression in Three Forms of Muscular Dystrophy. J Neuromuscul Dis. 2015 Sep 2;2(3):241-255. doi: 10.3233/JND-140066. PMID 26870665
- [Background] Carr, A. (2003). Adult Measures of Quality of Life: The Arthritis Impact Measurement Scales (AIMS/AIMS2), Disease Repercussion Profile (DRP), EuroQoL, Nottingham Health Profile (NHP), Patient Generated Index (PGI), Quality of Well-Being Scale (QWB), RAQoL, Short Form-36 (SF-36), Sickness Impact Profile (SIP), SIP-RA, and World Health Organization's Quality of Life Instruments (WHOQoL, WHOQoL-100, WHOQoL-Bref). Arthritis Care & Research, 49(S5), S113-S133. http://doi.org/10.1002/art.11414
- [Background] Centers for Disease Control and Prevention (CDC). Prevalence of doctor-diagnosed arthritis and arthritis-attributable activity limitation--United States, 2010-2012. MMWR Morb Mortal Wkly Rep. 2013 Nov 8;62(44):869-73. PMID 24196662
- [Background] Cerulli C, Minganti C, De Santis C, Tranchita E, Quaranta F, Parisi A. Therapeutic horseback riding in breast cancer survivors: a pilot study. J Altern Complement Med. 2014 Aug;20(8):623-9. doi: 10.1089/acm.2014.0061. Epub 2014 Jun 25. PMID 24963599
- [Background] Chaparro LE, Furlan AD, Deshpande A, Mailis-Gagnon A, Atlas S, Turk DC. Opioids compared to placebo or other treatments for chronic low-back pain. Cochrane Database Syst Rev. 2013 Aug 27;2013(8):CD004959. doi: 10.1002/14651858.CD004959.pub4. PMID 23983011
- [Background] Cho SH, Kim JW, Kim SR, Cho BJ. Effects of horseback riding exercise therapy on hormone levels in elderly persons. J Phys Ther Sci. 2015 Jul;27(7):2271-3. doi: 10.1589/jpts.27.2271. Epub 2015 Jul 22. PMID 26311966
- [Background] Dawson, S., & Liddicoat, K. (2009). "Camp Gives Me Hope": Exploring the Therapeutic Use of Community for Adults with Cerebral Palsy. Therapeutic Recreation Journal, 43(4), 9-24.
- [Background] de Araujo TB, de Oliveira RJ, Martins WR, de Moura Pereira M, Copetti F, Safons MP. Effects of hippotherapy on mobility, strength and balance in elderly. Arch Gerontol Geriatr. 2013 May-Jun;56(3):478-81. doi: 10.1016/j.archger.2012.12.007. Epub 2013 Jan 3. PMID 23290005
- [Background] Debuse D, Gibb C, Chandler C. Effects of hippotherapy on people with cerebral palsy from the users' perspective: a qualitative study. Physiother Theory Pract. 2009 Apr;25(3):174-92. doi: 10.1080/09593980902776662. PMID 19384737
- [Background] Duclos ME, Roualdes O, Cararo R, Rousseau JC, Roger T, Hartmann DJ. Significance of the serum CTX-II level in an osteoarthritis animal model: a 5-month longitudinal study. Osteoarthritis Cartilage. 2010 Nov;18(11):1467-76. doi: 10.1016/j.joca.2010.07.007. PMID 21056352
- [Background] Engel GL. The need for a new medical model: a challenge for biomedicine. Science. 1977 Apr 8;196(4286):129-36. doi: 10.1126/science.847460.
- [Background] Farias-Tomaszewski, S., Jenkins, S. R., & Keller, J. (2001). An evaluation of therapeutic horseback riding programs for adults with physical impairmnets. Therapeutic Recreation Journal, 35(3), 250.
- [Background] Fazio E, Medica P, Cravana C, Ferlazzo A. Hypothalamic-pituitary-adrenal axis responses of horses to therapeutic riding program: effects of different riders. Physiol Behav. 2013 Jun 13;118:138-43. doi: 10.1016/j.physbeh.2013.05.009. Epub 2013 May 15. PMID 23684906
- [Background] Felson DT, Lohmander LS. Whither osteoarthritis biomarkers? Osteoarthritis Cartilage. 2009 Apr;17(4):419-22. doi: 10.1016/j.joca.2009.02.004. Epub 2009 Feb 23. No abstract available. PMID 19248750
- [Background] Fernandes L, Hagen KB, Bijlsma JW, Andreassen O, Christensen P, Conaghan PG, Doherty M, Geenen R, Hammond A, Kjeken I, Lohmander LS, Lund H, Mallen CD, Nava T, Oliver S, Pavelka K, Pitsillidou I, da Silva JA, de la Torre J, Zanoli G, Vliet Vlieland TP; European League Against Rheumatism (EULAR). EULAR recommendations for the non-pharmacological core management of hip and knee osteoarthritis. Ann Rheum Dis. 2013 Jul;72(7):1125-35. doi: 10.1136/annrheumdis-2012-202745. Epub 2013 Apr 17. PMID 23595142
- [Background] Fieseler G, Molitor T, Irlenbusch L, Delank KS, Laudner KG, Hermassi S, Schwesig R. Intrarater reliability of goniometry and hand-held dynamometry for shoulder and elbow examinations in female team handball athletes and asymptomatic volunteers. Arch Orthop Trauma Surg. 2015 Dec;135(12):1719-26. doi: 10.1007/s00402-015-2331-6. Epub 2015 Sep 19. PMID 26386839
- [Background] Frevel D, Maurer M. Internet-based home training is capable to improve balance in multiple sclerosis: a randomized controlled trial. Eur J Phys Rehabil Med. 2015 Feb;51(1):23-30. Epub 2014 Apr 23. PMID 24755773
- [Background] George SZ, Wallace MR, Wu SS, Moser MW, Wright TW, Farmer KW, Borsa PA, Parr JJ, Greenfield WH 3rd, Dai Y, Li H, Fillingim RB. Biopsychosocial influence on shoulder pain: risk subgroups translated across preclinical and clinical prospective cohorts. Pain. 2015 Jan;156(1):148-156. doi: 10.1016/j.pain.0000000000000012. PMID 25599310
- [Background] Hakanson M, Moller M, Lindstrom I, Mattsson B. The horse as the healer-a study of riding in patients with back pain. J Bodyw Mov Ther. 2009 Jan;13(1):43-52. doi: 10.1016/j.jbmt.2007.06.002. Epub 2007 Aug 24. PMID 19118792
- [Background] Hammer A, Nilsagard Y, Forsberg A, Pepa H, Skargren E, Oberg B. Evaluation of therapeutic riding (Sweden)/hippotherapy (United States). A single-subject experimental design study replicated in eleven patients with multiple sclerosis. Physiother Theory Pract. 2005 Jan-Mar;21(1):51-77. doi: 10.1080/09593980590911525. PMID 16385943
- [Background] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Background] Homnick DN, Henning KM, Swain CV, Homnick TD. Effect of therapeutic horseback riding on balance in community-dwelling older adults with balance deficits. J Altern Complement Med. 2013 Jul;19(7):622-6. doi: 10.1089/acm.2012.0642. Epub 2013 Jan 29. PMID 23360659
- [Background] Homnick TD, Henning KM, Swain CV, Homnick DN. The effect of therapeutic horseback riding on balance in community-dwelling older adults: a pilot study. J Appl Gerontol. 2015 Feb;34(1):118-26. doi: 10.1177/0733464812467398. Epub 2012 Nov 28. PMID 25548091
- [Background] Hughes DC, Wallace MA, Baar K. Effects of aging, exercise, and disease on force transfer in skeletal muscle. Am J Physiol Endocrinol Metab. 2015 Jul 1;309(1):E1-E10. doi: 10.1152/ajpendo.00095.2015. Epub 2015 May 12. PMID 25968577
- [Background] Lee S, Lee D, Park J. Effects of the Indoor Horseback Riding Exercise on Electromyographic Activity and Balance in One-leg Standing. J Phys Ther Sci. 2014 Sep;26(9):1445-7. doi: 10.1589/jpts.26.1445. Epub 2014 Sep 17. PMID 25276033
- [Background] Karjalainen K, Malmivaara A, van Tulder M, Roine R, Jauhiainen M, Hurri H, Koes B. Multidisciplinary biopsychosocial rehabilitation for subacute low back pain in working-age adults: a systematic review within the framework of the Cochrane Collaboration Back Review Group. Spine (Phila Pa 1976). 2001 Feb 1;26(3):262-9. doi: 10.1097/00007632-200102010-00011. PMID 11224862
- [Background] Keren O, Reznik J, Groswasser Z. Combined motor disturbances following severe traumatic brain injury: an integrative long-term treatment approach. Brain Inj. 2001 Jul;15(7):633-8. doi: 10.1080/02699050010009568. PMID 11429091
- [Background] Kim HS, Lee CW, Lee IS. Comparison between the Effects of Horseback Riding Exercise and Trunk Stability Exercise on the Balance of Normal Adults. J Phys Ther Sci. 2014 Sep;26(9):1325-7. doi: 10.1589/jpts.26.1325. Epub 2014 Sep 17. PMID 25276009
- [Background] Kim SG, Lee CW. The effects of hippotherapy on elderly persons' static balance and gait. J Phys Ther Sci. 2014 Jan;26(1):25-7. doi: 10.1589/jpts.26.25. Epub 2014 Feb 6. PMID 24567669
- [Background] Kim SR, Cho SH, Kim JW, Lee HC, Brienen M, Cho BJ. Effects of horseback riding exercise therapy on background electroencephalograms of elderly people. J Phys Ther Sci. 2015 Jul;27(7):2373-6. doi: 10.1589/jpts.27.2373. Epub 2015 Jul 22. PMID 26311985
- [Background] Kolber MJ, Hanney WJ. The reliability and concurrent validity of shoulder mobility measurements using a digital inclinometer and goniometer: a technical report. Int J Sports Phys Ther. 2012 Jun;7(3):306-13. PMID 22666645
- [Background] Lechner HE, Feldhaus S, Gudmundsen L, Hegemann D, Michel D, Zach GA, Knecht H. The short-term effect of hippotherapy on spasticity in patients with spinal cord injury. Spinal Cord. 2003 Sep;41(9):502-5. doi: 10.1038/sj.sc.3101492. PMID 12934090
- [Background] Lechner HE, Kakebeeke TH, Hegemann D, Baumberger M. The effect of hippotherapy on spasticity and on mental well-being of persons with spinal cord injury. Arch Phys Med Rehabil. 2007 Oct;88(10):1241-8. doi: 10.1016/j.apmr.2007.07.015. PMID 17908564
- [Background] Aliev RG, Gaziev RM, Abdulaev MA, Daitbegov MKh. [Experience with the treatment of acute pancreatitis with 5-fluorouracil in the light of late results]. Vestn Khir Im I I Grek. 1988 Jun;140(6):28-31. Russian. PMID 2464865
- [Background] Lee CW, Kim SG, An BW. The effects of horseback riding on body mass index and gait in obese women. J Phys Ther Sci. 2015 Apr;27(4):1169-71. doi: 10.1589/jpts.27.1169. Epub 2015 Apr 30. PMID 25995581
- [Background] Mackay-Lyons, M., Conway, C., & Roberts, W. (1988). Effects of therapeutic riding on patients with multiple sclerosis: a preliminary trial... horseback riding. Physiotherapy Canada, 40(2), 104-109.
- [Background] Menezes, K., Mendonça, Copetti, F., Wiest, M., Joner, Trevisan, C., Morais, & Silveira, A., Ferreira. (2013). Effect of hippotherapy on the postural stability of patients with multiple sclerosis: a preliminary study. Fisioterapia E Pesquisa, 20(1), 43-49.
- [Background] Milfont, T. L., & Duckitt, J. (2010). The environmental attitudes inventory: A valid and reliable measure to assess the structure of environmental attitudes. Journal of Environmental Psychology, 30(1), 80-94. http://doi.org/10.1016/j.jenvp.2009.09.001
- [Background] Munoz-Lasa S, Ferriero G, Valero R, Gomez-Muniz F, Rabini A, Varela E. Effect of therapeutic horseback riding on balance and gait of people with multiple sclerosis. G Ital Med Lav Ergon. 2011 Oct-Dec;33(4):462-7. PMID 22452106
- [Background] Nimer, J., & Lundahl, B. (2007). Animal-Assisted Therapy: A Meta-Analysis. Anthrozoos, 20(3), 225-238. http://doi.org/10.2752/089279307X224773
- [Background] Ratliffe, K. T., & Sanekane, C. (2009). Equine-assisted therapies: Complementary medicine or not? Australian Journal of Outdoor Education, 13(2), 33-43.
- [Background] Sager, A., Drache, M., Schaar, B., & Pöhlau, D. (2008). Hippotherapy for multiple sclerosis - Pilot study assessing effects on balance, spasticity, ability to walk and quality of life. Multiple Scerosis, 14(1), S151.
- [Background] Schaafsma FG, Whelan K, van der Beek AJ, van der Es-Lambeek LC, Ojajarvi A, Verbeek JH. Physical conditioning as part of a return to work strategy to reduce sickness absence for workers with back pain. Cochrane Database Syst Rev. 2013 Aug 30;2013(8):CD001822. doi: 10.1002/14651858.CD001822.pub3. PMID 23990391
- [Background] Selby A, Smith-Osborne A. A systematic review of effectiveness of complementary and adjunct therapies and interventions involving equines. Health Psychol. 2013 Apr;32(4):418-32. doi: 10.1037/a0029188. Epub 2012 Aug 13. PMID 22888815
- [Background] Silkwood-Sherer D, Warmbier H. Effects of hippotherapy on postural stability, in persons with multiple sclerosis: a pilot study. J Neurol Phys Ther. 2007 Jun;31(2):77-84. doi: 10.1097/NPT.0b013e31806769f7. PMID 17558361
- [Background] Boxem KV, Zundert JV, van Kleef M. Re: Staal JB, de Bie R, de Vet HC, et al. Injection therapy for subacute and chronic low-back pain. Cochrane Database Syst Rev 2008:CD001824. Spine (Phila Pa 1976). 2009 Jul 1;34(15):1628-9; author reply 1629. doi: 10.1097/BRS.0b013e3181aa1ffa. No abstract available. PMID 19564780
- [Background] Sunwoo H, Chang WH, Kwon JY, Kim TW, Lee JY, Kim YH. Hippotherapy in adult patients with chronic brain disorders: a pilot study. Ann Rehabil Med. 2012 Dec;36(6):756-61. doi: 10.5535/arm.2012.36.6.756. Epub 2012 Dec 28. PMID 23342306
- [Background] Tseng SH, Chen HC, Tam KW. Systematic review and meta-analysis of the effect of equine assisted activities and therapies on gross motor outcome in children with cerebral palsy. Disabil Rehabil. 2013 Jan;35(2):89-99. doi: 10.3109/09638288.2012.687033. Epub 2012 May 26. PMID 22630812
- [Background] Global Recommendations on Physical Activity for Health. Geneva: World Health Organization; 2010. Available from http://www.ncbi.nlm.nih.gov/books/NBK305057/ PMID 26180873
- [Background] Yorke, J., Adams, C., & Coady, N. (2008). Therapeutic value of equine-human bonding in recovery from trauma. ANTHROZOOS, 21(1), 17-30.
- See also: Arthritis Impact Measurement Scale 2 — http://www.rheumatology.org/I-Am-A/Rheumatologist/Research/Clinician-Researchers/Arthritis-Impact-Measurement-Scales-AIMS
- See also: Range of Joint Motion Evaluation Chart — https://www.google.com/webhp?sourceid=chrome-instant&rlz=1C1AVNE_enUS621US621&ion=1&espv=2&ie=UTF-8#q=range+of+joint+motion+evaluation+chart